CLINICAL TRIAL: NCT01332045
Title: Continuous Saphenous Nerve Block (Adductor Channel) and Local Infiltration Analgesia (LIA) for Total Knee Arthroplasty
Brief Title: Continuous Saphenous Nerve Block for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henning Lykke Andersen (Other)
Responsible Party: Sponsor-Investigator, Henning Lykke Andersen, Consultant, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-3-2010-124
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline boluses in nerve catheter (Sham Comparator): A nerve catheter will be placed in the adductor canal using saline instead of Ropivacaine for intermittent boluses.
  Interventions: Procedure: Saline boluses in nerve catheter
- Continuous saphenous nerve block (Active Comparator): Postoperative intermittent boluses of 15 Ml Ropivacaine 7,5 mg/Ml every 12 hours for three days
  Interventions: Procedure: continuous saphenous nerve block

INTERVENTIONS:
Procedure: continuous saphenous nerve block — Postoperative intermittent boluses of 15 Ml Ropivacaine 7,5 mg/Ml every 12 hours for three days
  Arms: Continuous saphenous nerve block
Procedure: Saline boluses in nerve catheter — A nerve catheter will be placed in the adductor canal using saline instead of Ropivacaine for intermittent boluses.
  Arms: Saline boluses in nerve catheter

SUMMARY:
Our study will compare the use of continuous saphenous nerve block performed at the adductor canal in addition to Local Infiltration Analgesia (LIA) versus a Sham block in addition to LIA for total knee replacement. The investigators hypothesize that the saphenous nerve block performed at the level of the adductor canal in addition to LIA provides better pain relief than the LIA alone without significantly compromising muscle strength and physiotherapy, enabling patients to mobilize early with reduced opioid consumption and les side effects.

The investigators will enroll a total of 40 patients (20 patients will receive continuous saphenous nerve block in addition to LIA and 20 will receive the sham block and LIA). Until discharge, the investigators will record patients' pain scores, opioid consumption, side effects and physical therapy progress.

If our study proves that the continuous saphenous nerve block in addition to LIA can effectively reduce postoperative pain scores to an acceptable level with better physical therapy progress and less opioid consumption, it could be seen as a more attractive alternative to LIA alone or other traditionally used methods of postoperative pain control that compromises muscle strength and physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age: 40-75
* Unilateral TKA
* Use of Spinal anesthesia

Exclusion Criteria:

* Allergy to any of the study medications
* Intolerance to morphine
* Contraindication to a spinal anesthetic
* Intraoperative use of any volatile anesthetic
* Chronic opioid use
* ASA Class 4-5
* Rheumatoid arthritis or Diabetes mellitus with neuropathy
* Liver or kidney failure
* BMI above 40
* Severe COPD

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pain scores | 3 days postoperative
  VAS pain scores

SECONDARY OUTCOMES:
Opioid consumption | 3 days postoperative
physical therapy progress | 3 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Henning L. Andersen, M.D., Principal Investigator — Frederiksberg Hospital; Dusanka Zaric, M.D., Ph.d., Study Director — Frederiksberg Hospital.
Locations (1):
- Anaestesiafdelingen, Frederiksberg Hospital, Frederiksberg, Denmark

REFERENCES:
- [Derived] Andersen HL, Gyrn J, Moller L, Christensen B, Zaric D. Continuous saphenous nerve block as supplement to single-dose local infiltration analgesia for postoperative pain management after total knee arthroplasty. Reg Anesth Pain Med. 2013 Mar-Apr;38(2):106-11. doi: 10.1097/AAP.0b013e31827900a9. PMID 23222363
- See also: Related Info — http://www.frederiksberghospital.dk